CLINICAL TRIAL: NCT01496287
Title: Tympanostomy Tube Placement in Children in the Office (Inova Study)
Acronym: Inova
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005027
Record Dates: First submitted 2011-12-16; First posted 2011-12-21 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tube placement group (Experimental)
  Interventions: Device: Tube Delivery System (TDS)

INTERVENTIONS:
Device: Tube Delivery System (TDS) — Placement of tympanostomy tube by the Acclarent tympanostomy tube delivery system under local anesthesia in an office/clinic setting
  Other Names: Tula TDS

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Acclarent Tula TDS for the placement of tympanostomy tubes under local anesthesia in an office/clinic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo tympanostomy tube insertion
2. At least 6 months old and younger than 22 years old
3. Behavioral capacity and cooperative temperament to undergo an awake procedure (based on physician judgement)
4. No history of sensitivity or reaction to anesthesia chosen for the procedure

Exclusion Criteria:

1. Pregnant or lactating females
2. Significantly atrophic, bimeric, or completely atelectatic tympanic membrane
3. Otitis externa
4. Lacerations or abrasions to the external auditory canal or damaged or denuded skin in the auditory canal
5. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane
6. Electrically sensitive subjects and subjects with electrically sensitive support systems (pacemakers, defibrillators, etc.)
7. Anatomy that precludes sufficient visualization of and access to the tympanic membrane
8. Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob W Zeiders, M.D., Principal Investigator — South Coast Ear, Nose & Throat
Locations (1):
- South Coast Ear, Nose & Throat, Port Saint Lucie, Florida, United States

REFERENCES:
- [Derived] Zeiders JW, Syms CA, Mitskavich MT, Yen DM, Harfe DT, Shields RD, Lanier BJ, Gould AR, Mouzakes J, Elliott CL. Tympanostomy tube placement in awake, unrestrained pediatric patients: A prospective, multicenter study. Int J Pediatr Otorhinolaryngol. 2015 Dec;79(12):2416-23. doi: 10.1016/j.ijporl.2015.11.003. Epub 2015 Nov 10. PMID 26611339
- [Derived] Cohen LL, Martin SR, Gamwell KL, McCarty C, Shih SW. Behavioral techniques to optimize success of in-office pediatric tympanostomy tube placement without sedation. Int J Pediatr Otorhinolaryngol. 2015 Dec;79(12):2170-3. doi: 10.1016/j.ijporl.2015.09.041. Epub 2015 Oct 8. PMID 26514928

RESULTS

PARTICIPANT FLOW:
Groups:
- Tube Placement Group: Tube Delivery System (Tula): Placement of tympanostomy tube by the Acclarent tympanostomy tube delivery system following delivery of anesthetic with Acclarent iontophoresis device
Period: Overall Study
Arm/Group | Tube Placement Group
Started | 70
Completed | 64
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Incomplete anesthesia | 5

BASELINE CHARACTERISTICS:
Groups:
- Tube Placement Group: Tube Delivery System (Tula): Placement of tympanostomy tube by the Acclarent tympanostomy tube delivery system under local anesthesia in an office/clinic setting
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  African American or Black | 5
  Asian | 1
  White | 47
  Other or Unknown | 17
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural, Serious, and Device-Related Adverse Events
Description: Adverse events which are procedural, serious, and device-related.
Time Frame: procedure up to 2 weeks post procedure
Measure: Number; unit: participants
Groups:
- Tube Placement Group: Tube Delivery System (Tula): Placement of tympanostomy tube by the tympanostomy tube delivery system under local anesthesia in an office/clinic setting
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 70
participants | 0

2. Primary Outcome: Device Success
Description: Device Success is defined as the successful delivery of the tympanostomy tube (TT) across the tympanic membrane (TM) using the Tube Delivery System(TDS). Device Success will be evaluated on a per device basis.
Time Frame: Day 0 (day of procedure)
Population: Analysis population includes subjects who had completed the local anesthesia procedure (iontophoresis) and in which a TDS tube delivery device was attempted.
Measure: Number; unit: devices
Units Other Than Participants: devices
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 65
Number analyzed (devices) | 128
devices | 114

3. Secondary Outcome: Procedure Success
Description: Procedure Success is defined as the successful placement of any tympanostomy tube in all enrolled ears in a given subject. Procedure Success is determined on a per subject basis.
Time Frame: Day 0 (day of procedure)
Measure: Number; unit: participants
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 70
participants | 63

4. Secondary Outcome: Procedure Tolerability
Description: Procedure Tolerability is defined as the proportion of subjects reporting the procedure as tolerable, where tolerable is defined as a score of 0 through 3, using the Wong-Baker FACES pain scale.The Wong-Baker FACES pain scoring system is a scale of 0 to 5, where 0 means 'no hurt', 1 = 'hurts a little bit', 2 = 'hurts little more', 3 = 'hurts even more', 4 = 'hurts whole lot' and 5 = 'hurts worst'. Procedure Tolerability will be determined on a per patient basis, with the patient's score being the average of the scores for the left and right ear if both ears are successfully treated with the Tube Delivery System.
  "Tolerability" was defined as an average post-procedure pain score (of treated ears) <= "3"
Time Frame: Day 0 (day of procedure)
Measure: Number; unit: participants
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 64
participants | 59

5. Secondary Outcome: Tube Retention
Description: Tube retention is the presence of a tympanostomy tube placed successfully by the Tula TDS device across the tympanic membrane at the two-week follow-up visit.
Time Frame: 2 weeks post procedure
Population: Only 62 of the initial 70 subjects achieved procedure success, and were present for 2 week follow-up assessment with Tula tube in situ, such that tube retention could be measured.
Measure: Number; unit: ears
Units Other Than Participants: ears
Arm/Group | Tube Placement Group
Number analyzed (Participants) | 62
Number analyzed (ears) | 112
ears | 111

ADVERSE EVENTS:
Time Frame: procedure through 2 weeks post-procedure
Arm/Group | Tube Placement Group
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 3/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tube Placement Group (N=70)
occluded tube (Ear and labyrinth disorders) | 2 (2)
otalgia (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days